CLINICAL TRIAL: NCT01919632
Title: MOVING - Einfluß Eines Lebensstilprogramms Auf Gefaeßzustand, Metabolisches Risikoprofil Und Leistungsfaehigkeit (MOVING - Influence of a Lifestyle Intervention Program on Vascular Condition, Metabolic Risk Profile and Physical Performance)
Brief Title: MOVING - MOtiVation, INtervention and Vascular chanGe
Acronym: MOVING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Moving - ab jetzt gesund GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2555/09
Record Dates: First submitted 2013-07-05; First posted 2013-08-09 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Endothelial Function (Reactive Hyperemia)
Keywords: lifestyle; physical activity; endothelial function; cardiovascular; occupational; prevention
MeSH Terms: conditions — Hyperemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle (Experimental): The initial stage of the program consists of a health-behavior seminar and six weeks (twice a week for 90 minutes) of supervised endurance exercise (i.e. (?) jogging, nordic walking, cycling or swimming) in groups. In the second phase of the program, the participants receive a recommendation to continue exercise regularly unsupervised for one year, and receive monthly supervised exercise training sessions.
  Interventions: Behavioral: health-behavior seminar and endurance exercise

INTERVENTIONS:
Behavioral: health-behavior seminar and endurance exercise — The initial stage of the program consists of a health-behavior seminar and six weeks (twice a week for 90 minutes) of supervised endurance exercise (i.e. jogging, nordic walking, cycling or swimming) in groups. In the second phase of the program, the participants receive a recommendation to continue exercise regularly unsupervised for one year, and receive monthly supervised exercise training sessions.

SUMMARY:
Background: The impact of demographic changes on workplace has increased the importance of effective occupational preventive health programs. The primary goal of these programs is the improvement of overall health status (and therefore increase productivity and decrease healthcare costs) of the increasingly older workforce through positive lifestyle behavior change.

A one- year preventive health behavior-change program for the employees of the company British Petrol (BP) shall be scientifically evaluated. The initial stage of the program consists of a health-behavior seminar and six weeks (twice a week for 90 minutes) of supervised endurance exercise (i.e. jogging, nordic walking, cycling or swimming) in groups. In the second phase of the program, the participants receive a recommendation to continue exercise regularly unsupervised for one year, and receive monthly supervised exercise training sessions. Clinical check-ups are performed at baseline (V1) at three months (V2) and at 12 months (V3).

DETAILED DESCRIPTION:
The study will investigate the effect of one year of participation in a lifestyle- intervention- program on the participants' metabolic risk profile, exercise capacity and vascular health. A primary focus is on the endothelium, because poor endothelial health is a risk factor and prognostic indicator of atherosclerosis and cardiovascular events.

Hypothesis: One year of participation in endurance exercise (twice a week for 90 minutes) may positively influence endothelial health (RHI)

The primary aim:

change in endothelial function (reactive hyperemia index (RHI)) after one year.

Secondary aims:

Changes in other vascular parameters (AI: augmentation index, CAVI: Cardio ankle vascular index, ABI: ankle brachial index ), changes in anthropometric, inflammatory and metabolic parameters, exercise capacity (Watt/kg), physical activity, and health related quality of life (HRQoL).

ELIGIBILITY:
Inclusion Criteria:

* Employees of the company British Petrol (BP) in Lingen, Germany
* men and woman of all age
* approval for being able to participate in physical activity
* existing, written agreement to study-participation with prior, detailed education

Exclusion Criteria:

* Acute or chronic disease of any kind, which does not allow participation in physical activity (missing approval of being able to participate in physical activity)
* Incompetent patient, who is not able to understand character, meaning and consequences of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in RHI (Reactive Hyperemia Index) | after 0 months (V1), 3 months (V2), 12 months (V3)
  endothelial function

SECONDARY OUTCOMES:
Exercise capacity (Watt/kg) | after 0 month (V1) and after 12 month (V3)
  Changes from baseline in exercise capacity (Watt/kg) at 12 month
CAVI (Cardio ankle vascular index) | after 0 months (V1), 3 months (V2), 12 months (V3)
  Vascular function: Change from baseline in CAVI (Cardio ankle vascular index) at 12 month
Anthropometric parameters (see description) | after 0 months (V1), 3 months (V2), 12 months (V3)
  Changes from Baseline in systolic/diastolic blood pressure, weight, body-fat and waist-circumference at 12 month
Inflammatory and metabolic parameters from blood samples (see description) | after 0 month (V1), 3 month (V2), 12 month (V3)
  Change from baseline in blood glucose, HbA1c, total cholesterol, HDL, LDL, triglycerides (metabolic parameters) and C-reactive protein (inflammatory parameters)at 12 month
Health related quality of life (HRQoL) | after 0 month (V1) and 12 month (V3)
  questionnaire
AI (Augmentation Index) | after 0 month, 3 month, 12 month
  Vascular function: Change from baseline in AI (Augmentation Index) at 12 month
ABI (Ankle-Brachial-Index) | after 0 month, 3 month, 12 month
  Vascular function: Change from baseline in ABI (Ankle-Brachial-Index)at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, Prof., Study Chair — Klinikum rechts der Isar, Department of Prevention and Sports medicine, Technische Universität München
Locations (2):
- Germany (2):
  - Klinikum rechts der Isar, Technische Universität München, Munich, Bavaria
  - BP Lingen, Lingen, Emsland

REFERENCES:
- [Derived] Schaller N, Blume K, Hornig M, Senker L, Wolfarth B, Schuster T, Halle M, Esefeld K; MOVING (MOtiVation, INtervention and Vascular chanGe) study group. Occupational life-style programme over 12 months and changes of metabolic risk profile, vascular function, and physical fitness in blue-collar workers. J Occup Med Toxicol. 2023 Mar 22;18(1):4. doi: 10.1186/s12995-023-00370-w. PMID 36949505